CLINICAL TRIAL: NCT02613988
Title: Early Response Assessment Using on 3T Advanced MR Imaging as Predictor of Long-term Treatment Response in Newly Diagnosed Glioblastomas
Brief Title: Advanced MR Imaging as Predictor of Treatment Response in Newly Diagnosed Glioblastomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Sung Kim, Associate Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AsanMCHSKim_01
Record Dates: First submitted 2015-11-18; First posted 2015-11-25 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Adult Glioblastoma
Keywords: Glioblastoma; MRI; standard treatment
MeSH Terms: conditions — Glioblastoma | interventions — Diffusion Magnetic Resonance Imaging; Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR imaging and standard treatment (Other): Patients with glioblastoma undergo 3-Tesla magnetic resonance imaging to measure tumor protein content (using CEST-MRI), cellularity (using DW-MRI), and perfusion (using DCE-MRI and DSC-MRI with IV administration of gadolinium-containing contrast agent) at pre-CCRT; 4 weeks after completion of the CCRT; and every 2 or 3 months during the adjuvant temozolomide therapy.
  Interventions: Device: 3 Tesla magnetic resonance imaging; Device: Chemical exchange saturation transfer MRI; Device: Diffusion weighted MRI; Device: Dynamic susceptibility contrast MRI

INTERVENTIONS:
Device: 3 Tesla magnetic resonance imaging — High resolution structural imaging (contrast-enhanced T1-weighted image, T2-weighted image, Fluid-attenuated inversion recovery)
Device: Chemical exchange saturation transfer MRI — Amide proton transfer-weighted image
Device: Diffusion weighted MRI — diffusion-weighted image with b value 0, 1000, and 3000
Device: Dynamic susceptibility contrast MRI — dual echo EPI sequence

SUMMARY:
This clinical trial studies advanced MR imaging techniques in measuring early response of standard treatment may become predictors of long-term treatment response in patients with newly diagnosed glioblastomas.

DETAILED DESCRIPTION:
The standard care of patients with glioblastoma is concomitant chemoradiation and adjuvant temozolomide. Allowing for assessment of tumor therapy prior to treatment completion is important to select patients most likely to benefit from alternative treatment option. Multimodal advanced MR imaging- contrast-enhanced T1 weighted imaging, diffusion-weighted imaging, chemical exchange saturation transfer imaging, and perfusion imaging on 3T enables quantitative assessment of treatment response. Quantifying changes in advanced MR imaging techniques would allow predict outcome for early and long-term treatment response and survival in glioblastomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiologically and histologically confirmed diagnosis of newly diagnosed glioblastoma
* Patients must have measurable disease, defined as evident tumors with gadolinium enhancement on MRI that is measurable in at least one diameter
* Life expectancy of greater than 3 months
* Patients scheduled for standard therapy (6 weeks radiation treatment (RT) ~ 60 Gy, plus temozolomide 75 mg/m^2 during 6 week RT, and followed routine monthly temozolomide therapy)
* Ability to understand and the willingness to sign a written informed consent document; all patients, or their legal guardians, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines

Exclusion Criteria:

* Patients who underwent complete resection
* Patients with no evidence of measurable disease after surgery
* Patients who have had chemotherapy or radiotherapy
* Patients who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, electronic infusion pumps, etc), because such devices may be displaced or malfunction
* Patients who are pregnant or breast feeding; urine pregnancy test will be performed on women of child bearing potential
* For patients who have undergone surgical resection prior to joining the study, in whom baseline magnetic resonance (MR) images exhibit enough signal degradation (due to susceptibility artifact in the region of the surgical bed) such that the data are uninterpretable will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of Response Rate | 6 month
  The response was determined by a modification of the RANO criteria that combined the image assessment, neurologic evaluation and assessment of steroid use. Clinical and radiologic assessments were carried out at pre-CCRT; 4 weeks after completion of the CCRT; and every 2 or 3 months during the adjuvant TMZ therapy. Complete Response (CR) was defined as complete disappearance on MR of all enhancing tumor; Partial Response (PR) was defined as greater than or equal to 50% reduction in tumor size on MR by bi-dimensional measurement; Pseudoprogression was defined when there was a decrease or stabilization of the contrast-enhancing lesions for a minimum of six months and combined with no change in treatment/ or a increase in contrast-enhancing lesion on the first subsequent follow-up MR image, as long as it stabilized on the second follow-up and there was no need for treatment change. Responder = CR+PR+Pseudoprogression, Non-responder = Progression.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | On-study date to lesser of date of progression or date of death from any cause (assessed at 6 months)
  Estimated probable duration of life without disease progression, from on-study date to earlier of progression date or date of death from any cause, using the Kaplan-Meier method with censoring. Disease progression is defined under Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as >=20% increase in sum of longest diameters (LD) of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Quantitative changes to tumor protein content and tumor acidosis | Baseline imaging within 4 weeks after surgery and 4 weeks after completion of CCRT
  Amide proton transfer asymmetry (APTasym, %) from Chemical Exchange Saturation Transfer (CEST) Amine proton transfer asymmetry (AmPTasym %) from CEST
Quantitative changes to tumor cellularity | Baseline imaging within 4 weeks after surgery and 4 weeks after completion of CCRT
  Apparent diffusion coefficient (ADC, mm2/s) from Diffusion weighted MRI
Quantitative changes to tumor perfusion using dynamic susceptibility contrast MRI | Baseline imaging within 4 weeks after surgery and 4 weeks after completion of CCRT
  Normalized Cerebral blood volume (CBV, %) from dynamic susceptibility contrast (DSC)-MRI
Quantitative changes to tumor perfusion using dynamic contrast enhancement MRI | Baseline imaging within 4 weeks after surgery and 4 weeks after completion of CCRT
  Initial area-under-the-curve (IAUC) from dynamic contrast enhancement (DCE)-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sung Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Galban CJ, Chenevert TL, Meyer CR, Tsien C, Lawrence TS, Hamstra DA, Junck L, Sundgren PC, Johnson TD, Galban S, Sebolt-Leopold JS, Rehemtulla A, Ross BD. Prospective analysis of parametric response map-derived MRI biomarkers: identification of early and distinct glioma response patterns not predicted by standard radiographic assessment. Clin Cancer Res. 2011 Jul 15;17(14):4751-60. doi: 10.1158/1078-0432.CCR-10-2098. Epub 2011 Apr 28. PMID 21527563
- [Background] Park JE, Kim HS, Goh MJ, Kim SJ, Kim JH. Pseudoprogression in Patients with Glioblastoma: Assessment by Using Volume-weighted Voxel-based Multiparametric Clustering of MR Imaging Data in an Independent Test Set. Radiology. 2015 Jun;275(3):792-802. doi: 10.1148/radiol.14141414. Epub 2015 Jan 21. PMID 25611736
- [Background] Park JE, Kim HS, Park KJ, Kim SJ, Kim JH, Smith SA. Pre- and Posttreatment Glioma: Comparison of Amide Proton Transfer Imaging with MR Spectroscopy for Biomarkers of Tumor Proliferation. Radiology. 2016 Feb;278(2):514-23. doi: 10.1148/radiol.2015142979. Epub 2015 Aug 19. PMID 26491847
- [Derived] Moon HH, Park JE, Kim N, Kim YH, Song SW, Hong CK, Kim JH, Kim HS. Prospective longitudinal analysis of imaging-based spatiotemporal tumor habitats in glioblastoma, IDH-wild type: implication in patient outcome using multiparametric physiologic MRI. BMC Cancer. 2024 Sep 27;24(1):1197. doi: 10.1186/s12885-024-12939-7. PMID 39334005